CLINICAL TRIAL: NCT01094249
Title: An Open-Label, Drug-Drug Interaction Study to Evaluate the Effect of Paliperidone Extended-Release on the Steady-State Pharmacokinetics of Valproic Acid in Clinically Stable Subjects With Schizophrenia, Bipolar I Disorder or Schizoaffective Disorder
Brief Title: A Drug Interaction Study of Valproic Acid and Paliperidone Extended-Release (ER) in Patients With Schizophrenia, Bipolar I Disorder, or Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR017029; R076477BIM1004 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-02-18; First posted 2010-03-26 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia; Bipolar Disorder; Psychotic Disorders
Keywords: Paliperidone ER; INVEGA; Divalproex sodium; Depakote ER; Valproic acid; Pharmacokinetics; R076477BIM1004
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): divalproex sodium ER/paliperidone ER Divalproex sodium ER (dose determined from the patients prescreening therapeutic dose) once daily from Day 1 through Day 7 and once daily in combination with paliperidone ER 12 mg from Day 8 through Day 12
  Interventions: Drug: divalproex sodium ER/paliperidone ER

INTERVENTIONS:
Drug: divalproex sodium ER/paliperidone ER — Divalproex sodium ER (dose determined from the patients prescreening therapeutic dose) once daily from Day 1 through Day 7 and once daily in combination with paliperidone ER 12 mg from Day 8 through Day 12

SUMMARY:
The purpose of this study is to evaluate the potential effect of multiple oral doses of an extended release formulation of paliperidone on the pharmacokinetics (blood levels) of valproic acid (VPA) in patients with schizophrenia, bipolar I disorder, or schizoaffective disorder.

DETAILED DESCRIPTION:
This is an open-label (patient will know the identity of the study drug they are taking) study in patients diagnosed with either schizophrenia, bipolar I disorder, or schizoaffective disorder who currently receive treatment with valproic acid, sodium valproate, or divalproex sodium. The primary purpose of the study is to determine the effect, if any, that multiple doses of paliperidone extended release (ER) tablets has on the pharmacokinetics (ie, blood levels) of valproic acid administered in the study as divalproex sodium extended release (ER). Divalproex sodium consists of a compound of sodium valproate and valproic acid in a 1:1 molar relationship in an enteric coated form. Approximately 16 patients will take part in the study. The study will last approximately 41 days and participation in this study will require a minimum of 5 overnight stays up to a maximum of 13 overnight stays during study drug treatment. The study will consist of a screening period that will occur up to 21 days before study treatment, a 13-day treatment period, and a posttreatment period that will include a follow-up visit 1 week after end-of-treatment procedures are performed. The purpose of the screening visit is to see patients meet all of the requirements to participate in the study. At the screening visit, after patients read and provide written informed consent acknowledging their willingness to participate in the study, the following procedures will be performed: 1) information regarding medical, psychiatric, and surgical history and medications currently taken will be collected, 2) a physical examination will be performed, 3) vital signs (blood pressure) and an electrocardiogram (ECG, a painless test to measure the electrical activity of the heart) will be assessed, 4) a blood sample for routine laboratory tests as well as to test for hepatitis B, hepatitis C, and human immunodeficiency virus (HIV) (and to check for pregnancy in women of child-bearing potential) will be collected, 5) a urine sample will be collected for routine laboratory testing including testing for drugs of abuse, and 6) an alcohol breath test will be performed. Patients who meet entry criteria for the study will be asked to check-in at the study clinic the evening before the first administration of study drug and will stay overnight at the clinic for at least 5 days or through Day 13 (approximately 2 weeks). During overnight stays at the clinic, patients will be required to eat and drink only the meals and beverages provided at the clinic. Patients will take each study drug orally (by mouth) in the following order on the days specified: divalproex sodium ER once daily for 7 days (Day 1 through Day 7) followed by divalproex sodium ER once daily in combination with paliperidone ER once daily for 7 days (ie, Days 8 through Day 12). During the study, patients will have blood samples taken from a vein in their arm using a needle (or flexible tube) at specified times during the study to determine the concentration of drugs in their blood. On Day 13 (or at the time of early withdrawal from the study) after the last blood sample for drug levels has been collected, patients will undergo end-of-study procedures that will include a physical examination, measurement of vital signs, and an ECG. A blood and urine sample for routine laboratory testing will also be collected during the end-of-study procedures to check the patients general health (and to check for pregnancy in women of child-bearing potential). After all end-of-study procedures have been completed, patients will leave the study clinic and return in about 1 week for a posttreatment follow-up visit where their overall general condition and the occurrence of any adverse events will be assessed. The primary objective of this study is to assess the potential effect of multiple doses of paliperidone ER tablets on the steady state pharmacokinetics of VPA. Steady state is achieved when drug concentrations in the blood are stable (ie, when the rate of drug absorption equals the rate of drug elimination in the body). Patients will also be monitored for safety from the time that they sign the informed consent form through to the end of the study (ie, posttreatment follow up visit). Safety will include monitoring adverse events, changes in clinical laboratory test results, ECG parameters, vital signs measurements, physical examination findings, the severity of the patients general condition, and concomitant medications (medications other than study drugs taken by patients) throughout the study period. All patients will receive a single oral (by mouth) daily dose of divalproex sodium ER (dose depended on the patients prescreening therapeutic dose) on Days 1 through 7 and divalproex sodium ER once daily in combination with one 12mg tablet of paliperidone ER once daily on Days 8 through 12. All study drugs are to be swallowed whole with water.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Is clinically stable with no psychiatric hospitalization or change in existing mood stabilizers, antipsychotic, or anti-manic drugs for 1 month before screening
* Taking valproate (valproic acid, sodium valproate, or divalproex sodium) for a minimum of 4 weeks before screening with a stable therapeutic dose for a minimum of 2 weeks and have confirmed therapeutic blood concentrations at screening
* If a woman, be postmenopausal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry and throughout the study
* If a man, agrees to use an adequate contraception method as deemed appropriate by the Investigator and to not donate sperm using the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Meet DSM-IV criteria for rapid cycling if primary diagnosis is bipolar I disorder
* DSM-IV diagnosis of alcohol or substance abuse with the exception of nicotine or caffeine dependence, within 12 months before screening
* Current suicidal ideation or violent tendencies at the time of screening
* History of neuroleptic malignant syndrome, any malignancy (with exception of basal cell carcinoma) within the past 5 years, any severe pre-existing gastrointestinal narrowing, or any history (or presence) of any cardiovascular, respiratory, neurologic, renal, hepatic, gastrointestinal, endocrine, hematologic, or immunologic disease
* moderate or severe tardive dyskinesia at the time of screening
* known allergy or intolerance of study drugs (ie, paliperidone, the parent compound risperidone, valproic acid, sodium valproate, or divalproex sodium) or any of the excipients of the formulations (eg, lactose)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the potential effect of multiple doses of paliperidone ER tablets on the steady state pharmacokinetics of VPA. | Blood samples collected at specified times on Days 4 through 13.

SECONDARY OUTCOMES:
To evaluate safety and tolerability of paliperidone ER coadministered with divalproex sodium ER | From time of screening (Day -21 up to Day -2) through the posttreatment follow-up visit 1 week after the end-of-study visit (Day 13 or time of early withdrawal from study)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- United States (3):
  - Kissimmee, Florida
  - Austin, Texas
  - Portsmount, Virginia

REFERENCES:
- See also: A Drug Interaction Study of Valproic Acid and Paliperidone Extended-Release (ER) in Patients with Schizophrenia, Bipolar I Disorder, or Schizoaffective Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=845&filename=CR017029_CSR.pdf